CLINICAL TRIAL: NCT06948370
Title: The PARADIGM-Q Study: Development and Evaluation of a Culturally Sensitive Problem- and AttributesbAsed DIabetes Self-Management Program for People With Type 2 Diabetes Residing in Qatar
Brief Title: Development and Evaluation of a Culturally Sensitive Structured Diabetes Self-Management Program for People With Type 2 Diabetes Residing in Qatar
Acronym: PARADIGM-Q
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ragae Dughmosh (Other)
Collaborators: Qatar National Research Fund (Other); Hamad Medical Corporation (Industry); Primary Health Care Corporation, Qatar (Other Government); Qatar University (Other)
Responsible Party: Sponsor-Investigator, Ragae Dughmosh, PhD Student, Qatar University
Organization: Qatar University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ARG02-0403-240132
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Self-management; Type 2 Diabetes Mellitus (T2DM); Diabetes Self-management
Keywords: Type 2 Diabetes Mellitus; Diabetes self-management; Quasi Experimental trial; systematic review and dose response meta-analysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study employing a parallel assignment model. Participants with Type 2 Diabetes Mellitus will be allocated to either the intervention group receiving the newly developed PARADIGM-Q diabetes self-management education program or the control group receiving the standard DESMOND program. The study aims to compare outcomes across these two groups without individual or health center randomization, using systematic allocation based on predefined inclusion criteria and institutional referral pathways."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARADIGM-Q Intervention Arm (Experimental): PARADIGM-Q Intervention Arm (Experimental):
  Participants in this arm will receive the PARADIGM-Q Diabetes Self-Management Education (DSME) program. This is a culturally sensitive, structured education intervention developed using the PARADIGM model and delivered through Case-Based Learning (CBL). The program consists of three weekly sessions (each lasting 3.5 hours) covering core self-management attributes: problem-solving, decision-making, taking action, resource utilization, and patient-provider relationships.
  Interventions: Behavioral: Intervention Name: PARADIGM-Q Diabetes Self-Management Education Program
- DESMOND Control Arm (Active Comparator): DESMOND Control Arm (Active Comparator) Participants in this arm will receive the DESMOND (Diabetes Education and Self-Management for Ongoing and Newly Diagnosed) program, which is the standard DSME program currently implemented in Qatar. It involves two group sessions (each lasting approximately 4 hours) and focuses on providing theoretical-based diabetes education for ongoing and newly diagnosed Type 2 Diabetes patients.
  Interventions: Behavioral: Control Arm (DESMOND): DESMOND Diabetes Self-Management Education Program

INTERVENTIONS:
Behavioral: Intervention Name: PARADIGM-Q Diabetes Self-Management Education Program — PARADIGM-Q Diabetes Self-Management Education Program This is a culturally sensitive, structured education intervention tailored for adults with Type 2 Diabetes in Qatar. Developed using the PARADIGM model and delivered through a Case-Based Learning (CBL) approach, the program comprises three weekly group sessions of 3.5 hours each. Each session targets key self-management attributes: problem-solving, decision-making, taking action, resource utilization, and patient-provider relationships. The program emphasizes real-life applicability, cultural relevance, and skill-building to support sustainable diabetes self-care.
  Arms: PARADIGM-Q Intervention Arm
Behavioral: Control Arm (DESMOND): DESMOND Diabetes Self-Management Education Program — The DESMOND Diabetes Self-Management Education Program is the standard diabetes education intervention currently offered to newly diagnosed patients with Type 2 Diabetes in Qatar. It is a UK-developed, theory-driven program delivered over two group sessions, each lasting approximately four hours. The program provides structured education on diabetes, lifestyle management, and risk reduction strategies. It does not incorporate case-based learning or cultural tailoring, distinguishing it from the experimental PARADIGM-Q intervention. DESMOND is used here as an active comparator to evaluate the added value of culturally sensitive, problem-based education.
  Arms: DESMOND Control Arm

SUMMARY:
This study is about helping people in Qatar who have Type 2 Diabetes take better care of their health. Diabetes is a common and growing problem in Qatar, and many people need more support and information to manage it well in their daily lives.

Right now, there is a program called DESMOND in Qatar, but it is only available in a few places and can be expensive to run. It also doesn't always work well in the long term. That's why we are creating a new diabetes education program called PARADIGM-Q. This program will be easier to access, more affordable, and designed to match the culture and needs of people living in Qatar.

The PARADIGM-Q program will teach people how to manage diabetes using real-life examples and group discussions. This method is called Case-Based Learning. It helps people understand their condition better and learn how to make good decisions about food, exercise, medication, and dealing with challenges.

The project will happen in two main phases:

Phase One: Understanding and Creating the Program

In the first part, we'll look at different ways of teaching about diabetes and see if a method called Case-Based Learning (CBL) works well. After that, we'll build a curriculum (a plan for teaching) based on the PARADIGM model. This curriculum, called the PARADIGM-Q program, will use the CBL method to teach. We'll also test this new program with a small group of diabetes educators and people with diabetes to make sure it works well. Their feedback will help me make the program even better.

Phase Two: Testing the Program

In the second part, we'll do a big study using a mix of people from different backgrounds in Qatar who have Type 2 Diabetes. we want to see if the PARADIGM-Q program is better than the program they already have (called DESMOND). we'll look the impact of our new program on different things like how much they know about diabetes, how active they are, their blood sugar levels (HbA1C), and their overall quality of life.

This study could lead to a new standard for diabetes education in Qatar and other countries in the region, helping more people live healthier lives with diabetes.

DETAILED DESCRIPTION:
This PhD research project aims to develop and evaluate a culturally sensitive Diabetes Self-Management Education (DSME) program, the PARADIGM-Q, specifically tailored for people with Type 2 Diabetes Mellitus (T2DM) residing in Qatar. With T2DM reaching epidemic levels globally and particulary among Qatar's population(1), there is an urgent need for effective DSME programs that are tailored to the country's needs. Current DSME programs, such as DESMOND-Qatar, have many limitations, including the fact that it is only available in two places, limiting access to many people who could benefit from diabetes education. Furthermore, the certification and recertification of DESMOND educators are rather costly, presenting financial barriers to the scaling up of this model; it is also limited in its long-term effectiveness(2), increasing the need for a sustainable and culturally appropriate solution to enable people with diabetes to self- manage their condition effectively. In this project, I will employ the locally developed PARADIGM model(3) framework to structure the new DSME interventions across two phases. In the initial phase, the focus is on developing a practical working curriculum using this model. This curriculum, named the PARADIGM-Q program, will incorporate the Case-Based Learning (CBL)(4) approach as its teaching delivery method. A systematic review and dose-response meta-analysis of relevant literature related to the optimal characteristics and duration of the program, followed by the development and piloting of the PARADIGM-Q curriculum. The curriculum will be refined through feedback obtained. The second phase involves evaluating the program's effectiveness through a Quasi-Experimental study, comparing it with Qatar's existing Diabetes Education Self-Management for Ongoing and Newly Diagnosed (DESMOND) program. The development of our local novel (PARADIGM-Q) will promote long-term effectiveness and patient adherence by combining the case-based Learning (CBL) approach with PARADIGM model. In addition, it will also emerge as a cost-effective alternative by establishing a central hub for training trainers within the Qatar health system, encompassing PHCC, HMC, Military Health Services, and private sectors. The primary research question is whether a culturally sensitive, case-based DSME program (PARADIGM-Q) can improve clinical and behavioral outcomes more effectively than existing models. This project has the potential to set a new standard for diabetes education in Qatar and the broader Gulf region, offering a scalable, sustainable intervention that aligns with local cultural practices and healthcare needs.

PROJECT STRUCTURE AND RESEARCH APPROACH

OBJECTIVES AND SIGNIFICANCE

Hypothesis:

The primary hypothesis is that implementing a culturally sensitive, case-based and attributes-based diabetes self-management education program (PARADIGM-Q) will significantly improve clinical outcomes, self-management behaviors, and quality of life for people with Type 2 Diabetes Mellitus (T2DM) when compared to the current DESMOND program.

Study Aim:

To Develop a culturally sensitive and well-structured Diabetes Self-Management Education (DSME) Program tailored specifically for individuals with Type 2 Diabetes residing in Qatar. This program will be developed based on the PARADIGM (Problem And attRibutes-bAsed DIabetes self-manaGeMent) model(3).

Objectives

1. To Create the curriculum for a culturally sensitive DSME program using Case-Based Learning (CBL) methodology, aligned with the PARADIGM model's core attributes, and tailored to Qatar's cultural variations.
2. Pilot study to validate a newly established DSME curriculum for feasibility, comprehensibility, relevance, and cultural sensitivity among diabetes educators and T2DM patients.
3. Effectiveness study to determine the impact of the PARADIGM-Q program on clinical outcomes, self-management behaviors, and quality of life compared to the DESMOND program using a robust quasi-experimental design.

METHODOLOGICAL APPROACHES

Type and classification of study:

Several research designs will be used for this study.

Phase One:

1. Systematic Review Objective: To examine the durability of standard diabetes self-management education program on glycosylated hemoglobin (HbA1c) levels over time, and to identify optimal DSME characteristics for glycemic control, forming the basis for the PARADIGM-Q curriculum.

   Methodology: Conduct a rigorous systematic review and dose response meta-analysis of data from existing studies of conventional DSME programs to gather evidence to determine the optimal duration of effect on glycemic control.

   Expected Outcome: Synthesize findings to inform on the current baseline before we develop and test our new culturally sensitive DSME program. Our study results will then be compared to results from the evidence synthesis on the durability of current programs on glycemic control.
2. Curriculum Formulation and Pilot Study Objective: Formulate a core-attributes, problem-based curriculum based on the PARADIGM model, And to collect feedback for refining the curriculum and ensuring it meets the educational and cultural needs of the Qatari population.

   Methodology

   Design:
   * A mixed methods study design will be used and will involve diabetes educators and participants with T2DM in a pilot study to validate the PARADIGM-Q curriculum.
   * Utilize focus group, pre-post assessments and semi-structured interviews with participants diagnosed with T2DM and diabetes educators to gather feedback on the curriculum's comprehensibility, relevance, and cultural sensitivity. Subsequently, refine curriculum components based on the insights obtained.

   Expected Outcome: A validated and culturally sensitive DSME program curriculum ready for implementation which will be called the PARADIGM-Q program.

   Sampling:
   * Technique: Non-probability quota sampling
   * Participants: 20 adults with Type 2 diabetes, divided by gender and language proficiency:

     * Male Arabic speakers
     * Female Arabic speakers
     * Male English speakers
     * Female English speakers This is especially relevant as the newly developed (PARADIGM-Q) program aims to address the needs of the multiethnic population residing in Qatar, encompassing individuals proficient in both Arabic and English languages.

   Curriculum Contents:

   PARADIGM-Q Program Structure:

   • Duration: The PARADIGM-Q program consists of three weekly sessions, each lasting three hours, designed to support effective diabetes management by integrating it into daily life routines.

   • Session Content:

   o Week 1: Problem Solving

   o Week 2: Decision Making and Taking Action.

   o Week 3: Resource Utilization, and Patient-Provider Relationships

   Educational Approach:

   • Case-Based Learning (CBL): Each session begins with a case scenario to stimulate discussion, problem-solving, and skills application.

   • Interactive Discussions: Each session closes with actionable strategies for taking learned skills back into your daily self-care routine.

   • Hands-on Demonstrations: The Facilitator (diabetes educators) aid by using demonstration tools to bridge these gaps.

   Data Collection and Analysis

   Quantitative Measures:

   • Pre- and Post-Program Assessments: Diabetes Knowledge Questionnaire (DKQ), Problem Areas in Diabetes (PAID) Scale, Ambulatory Glucose Profile (AGP) using a glucose sensor for two weeks pre and post the month of the intervention, and physical activity (monitored by smartwatches).

   Qualitative Measures:

   • Focus Groups: Conducted with T2D participants post-program about the curriculum's relevance, cultural sensitivity, and effectiveness of the educational approach.
   * Semi-Structured Interviews: Facilitators and participants will provide insights on session dynamics, instructional methods, and cultural appropriateness.

   Data Analysis:
   * Quantitative data will be analyzed for knowledge gains, stress reduction (PAID), and glycemic variability.
   * Qualitative data will undergo thematic analysis to derive insights into program relevance, effectiveness, and cultural fit.

   Expected Outcomes
   * A validated, culturally adapted DSME program (PARADIGM-Q) ready for large-scale implementation.
   * Qualitative and quantitative evidence of curriculum effectiveness and cultural resonance.

   Phase Two:

1- Controlled before-after Quasi-Experimental study Objective: Evaluate the effectiveness of the (PARADIGM-Q) program on various diabetes outcomes among people with T2DM in Qatar.

Expected Outcome: Empirical evidence on the effectiveness of our new culturally sensitive DSME program (PARADIGM-Q) compared to the existing program (DESMOND).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 65 years.
2. Diagnosed with Type 2 Diabetes Mellitus.
3. Most recent HbA1c ≥ 8% (within the last 6 months).
4. Fluent in Arabic and/or English.
5. Qatari and non-Qatari participants.
6. Able and willing to attend group-based education sessions.

Exclusion Criteria:

1. Diagnosed with any type of diabetes other than Type 2.
2. Pregnant women.
3. Presence of major diabetes complications (e.g., renal failure, severe retinopathy, blindness, stroke, heart failure, cancer).
4. Physical or mental disabilities that would hinder participation in education sessions.
5. Age below 18 or above 65 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) | Baseline, 3 months, 6 months, 9 months, 12 months post-intervention
  Measurement of HbA1c to assess long-term glycemic control.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life | Baseline and 3, 6, 9, 12 months post-intervention
  Evaluated using the Appraisal of Diabetes Scale (ADS)

CONTACTS AND LOCATIONS:
Overall Officials: Manal Musallam Othman, PhD, Principal Investigator — Hamad Medical Corporation

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, plans for sharing individual participant data (IPD) are under review and subject to ethical, institutional, and regulatory approvals. Data sharing will be considered based on the sensitivity of health information, participant confidentiality, and applicable data protection regulations. A final decision will be made in alignment with institutional policies and the requirements of the funding body.